CLINICAL TRIAL: NCT06086626
Title: A Multicenter, Single-arm, Open-label Study to Assess the Pharmacokinetics, Safety, and Tolerability of Cefiderocol in Hospitalized Pediatric Patients From Birth to < 3 Months of Age With Suspected or Confirmed Aerobic Gram-negative Bacterial Infections
Brief Title: A Study to Assess the Safety, Tolerability, and Pharmacokinetics of Cefiderocol in Hospitalized Neonates and Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Shionogi (Industry)
Responsible Party: Sponsor
Organization: Shionogi Inc. (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1904R2136
Record Dates: First submitted 2023-10-11; First posted 2023-10-17 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Gram-Negative Bacterial Infections
Keywords: Complicated urinary tract infection (cUTI); Complicated intra-abdominal infection (cIAI); Hospital-acquired bacterial pneumonia (HABP); Ventilator-associated (VABP); Bloodstream infection (BSI)/sepsis
MeSH Terms: conditions — Gram-Negative Bacterial Infections; Sepsis | interventions — Cefiderocol; Standard of Care

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Single-Dose Cefiderocol (Experimental): Participants will receive a single dose cefiderocol on Day 1, along with standard of care antibiotics
  Interventions: Drug: Cefiderocol; Drug: Standard of Care
- Multiple-Dose Cefiderocol (Experimental): Participants will receive cefiderocol every 8 hours for 5 to 14 days, along with standard of care antibiotics
  Interventions: Drug: Standard of Care

INTERVENTIONS:
Drug: Cefiderocol — Administered via intravenous (IV) infusion
  Other Names: S-649266
  Arms: Single-Dose Cefiderocol
Drug: Standard of Care — Antibiotics selected by the investigator based on the participant's symptoms, in accordance with local standards

SUMMARY:
The primary purpose of this study is to understand the pharmacokinetics (PK) of single and multiple doses of cefiderocol in children from birth to less than 3 months of age with suspected or confirmed aerobic Gram-negative bacterial infections.

ELIGIBILITY:
Eligibility Criteria: Key Inclusion Criteria:

1. Written informed consent has been provided by parent(s) or legally authorized representative(s) in accordance with local regulatory requirements
2. Hospitalized infants from birth to < 3 months (< 90 days) of age at the time written informed consent is provided. Enrollment of premature infants will not be restricted, but they must have a GA ≥ 26 weeks, PNA of 0 to 3 months, and weight of at least 1 kilogram (kg)
3. Require systemic IV antibiotic treatment for suspected or confirmed aerobic Gram-negative infections including, but not limited to, complicated urinary tract infection, complicated intra-abdominal infection, hospital-acquired/ ventilator-associated bacterial pneumonia, and BSI/sepsis
4. For the multiple-dose phase, within 72 hours of the start of potentially effective treatment with SOC antibiotics for the suspected or confirmed primary aerobic Gram-negative infection

Key Exclusion Criteria:

1. Documented history of any moderate or severe hypersensitivity or allergic reaction to any β-lactam antibiotic
2. Life expectancy of < 72 hours after enrollment
3. Urine output < 1.0 milliliter (mL)/kg/hour within the 24 hours prior to study drug administration on Day 1
4. Serum creatinine value greater than the maximum for GA and PNA shown below within the 24 hours prior to study drug administration on Day 1
5. Neonatal acute kidney injury (AKI), defined as a serum creatinine level greater than 1.5 milligrams per decilieter (mg/dL) (133 micromoles[μmol]/liter [L]) or an increase of 0.3 mg/dL (17 to 27 μmol/L) per day from a previous lower value
6. Acute kidney injury based on an increase in serum creatinine ≥ 0.3 mg/dL within 48 hours from an established baseline value
7. Any condition or circumstance that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data
8. Receiving renal replacement therapy
9. Received any other investigational medicinal product within 30 days of study drug administration
10. Receiving treatment with a vasopressor at Screening
11. Has a confirmed or strongly suspected infection at Screening with a pathogen known to be resistant to cefiderocol or only a Gram-positive pathogen or viral, fungal, or parasitic pathogen as the sole cause of infection
12. Anticipated need for antibacterial therapy longer than 14 days (example , osteomyelitis or endocarditis); this applies to both study treatment with cefiderocol, as well as adjunctive IV antibacterial treatment for suspected coinfection with Gram-positive organisms or multidrug resistant Gram-negative organisms
13. Suspected or confirmed central nervous system (CNS) infection, including suspected CNS infection who do not have a lumbar puncture (LP) but who are treated for potential CNS infection, evidence suggestive of CNS infection based on LP results (polymorphonuclear pleocytosis, hypoglycorrhachia, and increased protein concentration), regardless of culture results, LP with organisms on Gram stain or culture-positive cerebrospinal fluid

Note: Other protocol-defined Inclusion/Exclusion criteria may apply.

Max Age: 3 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2024-03-14 (Actual); Primary Completion 2025-03-31 (Actual); Study Completion 2025-03-31 (Actual)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) After a Single Dose of Cefiderocol | Up to 8 hours postdose
Cmax After a Minimum of 4 Doses of Cefiderocol | Up to 8 hours postdose
Area Under the Concentration-Time Curve Extrapolated From Time 0 to Infinity (AUC0-inf) After Single Dose of Cefiderocol | Up to 8 hours postdose
Area Under the Concentration-Time Curve Over the Dosing Interval (AUC0-†) After a Minimum of 4 Doses of Cefiderocol | Up to 3 hours
Terminal Elimination Half-Life (t1/2) After a Single Dose of Cefiderocol | Up to 8 hours postdose
Terminal Elimination Half-Life (t1/2) After a Minimum of 4 Doses of Cefiderocol | Up to 8 hours postdose

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) | Up to 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Shionogi
Locations (4):
- United States (2):
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Duke University, Durham, North Carolina
- Tygerberg Hospital, Cape Town, Western Cape, South Africa
- Chang Gung Memorial Hospital, Linkou Department of Pediatrics, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bradley JS, Orchiston E, Portsmouth S, Ariyasu M, Baba T, Katsube T, Makinde O. Pharmacokinetics, Safety and Tolerability of Single-dose or Multiple-dose Cefiderocol in Hospitalized Pediatric Patients Three Months to Less Than Eighteen Years Old With Infections Treated With Standard-of-care Antibiotics in the PEDI-CEFI Phase 2 Study. Pediatr Infect Dis J. 2025 Feb 1;44(2):136-142. doi: 10.1097/INF.0000000000004529. Epub 2024 Sep 4. PMID 39230271